CLINICAL TRIAL: NCT04007406
Title: DP13 - A Phase II Study in Patients With Primary Aldosteronism to Evaluate the Efficacy, Safety and Tolerability of DP13, Over an 8-week Treatment Period
Brief Title: DP13 - A Phase II Study in Patients With Primary Aldosteronism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Damian Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DP13C201
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Results first posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-10

CONDITIONS: Primary Aldosteronism
Keywords: Hyperaldosteronism
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 4 mg DP13 daily (Experimental): DP13 for 8 weeks
  Interventions: Drug: dexfadrostat phosphate
- 8 mg DP13 daily (Experimental): DP13 for 8 weeks
  Interventions: Drug: dexfadrostat phosphate
- 12 mg DP13 daily (Experimental): DP13 for 8 weeks
  Interventions: Drug: dexfadrostat phosphate

INTERVENTIONS:
Drug: dexfadrostat phosphate — DP13 systemic administration
  Other Names: DP13

SUMMARY:
The purpose of the present phase II study is to determine whether DP13 displays the clinical safety and efficacy profile to support further development in patients with primary aldosteronism.

DETAILED DESCRIPTION:
A phase II, multi-centre, randomized, parallel group, baseline-and withdrawal-controlled study in patients with primary aldosteronism to determine the dose-dependent efficacy, safety and tolerability of DP13 after a 2-week single-blind placebo run-in period followed by a randomized 8-week double-blind treatment period. After an additional single-blind, 2-week DP13 placebo withdrawal period, patients are switched to standard of care.

ELIGIBILITY:
Inclusion Criteria:

Patients with a guideline-recommended diagnosis of primary aldosteronism

Exclusion Criteria:

Patients with primary aldosteronism and

* hyperkalemia
* prolonged QT intervals
* refusal of special contraception measures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Mulatero, Prof, Principal Investigator — University of Torino, Torino, Italy
Locations (1):
- Ospedale Molinette, Torino, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited 'de novo' i.e., diagnosed with Primary Aldosteronism within 10 weeks of study entry or as 'recently diagnosed' i.e., diagnosed between 10 weeks and 1 year prior to study entry
Pre-assignment Details: Patient screening ARR and BP were reviewed and approved by the Eligibility Review Panel prior to study enrollment.
  A suppression test was required prior to study entry to confirm PA diagnosis. Patients had a 2-week placebo run-in prior to randomization.
Groups:
- 4 mg DP13: Patients receiving the low dose of dexfadrostat phosphate taken orally, once daily, in the morning before breakfast
- 8 mg DP13: Patients receiving the middle dose of dexfadrostat phosphate taken orally, once daily, in the morning before breakfast
- 12 mg DP13: Patients receiving the high dose of dexfadrostat phosphate taken orally, once daily, in the morning before breakfast
Period: Overall Study
Arm/Group | 4 mg DP13 | 8 mg DP13 | 12 mg DP13
Started | 10 | 12 | 13
Completed | 10 | 12 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 4 mg DP13; 8 mg DP13; 12 mg DP13: Baseline values were determined following 2 weeks of single-blind placebo run-in
- Total: Total of all reporting groups
Arm/Group | 4 mg DP13 | 8 mg DP13 | 12 mg DP13 | Total
Number analyzed (Participants) | 10 | 12 | 13 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 12 | 13 | 35
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 9
  Male | 7 | 9 | 10 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 9 | 11 | 13 | 33
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 7 | 7 | 9 | 23
  Netherlands | 0 | 1 | 1 | 2
  Switzerland | 3 | 4 | 3 | 10
Office systolic blood pressure (oSBP) [Mean (Standard Deviation); unit: mmHg] | 147 (14) | 148 (6) | 148 (14) | 148 (12)
Office diastolic blood pressure (oDBP) [Mean (Standard Deviation); unit: mmHg] | 90 (11) | 95 (9) | 92 (9) | 92 (10)
Aldosterone-to-renin ratio (ARR) [Median (Inter-Quartile Range); unit: ng*L/dL*mU] | 21.4 [6.8 to 28.9] | 7.2 [2.9 to 17.5] | 17.8 [9.0 to 25.2] | 15.3 [5.3 to 25.9]
24-hour ambulatory systolic blood pressure (aSBP) [Mean (Standard Deviation); unit: mmHg] | 137 (16) | 145 (14) | 145 (13) | 143 (14)
24-hour ambulatory diastolic blood pressure (aDBP) [Mean (Standard Deviation); unit: mmHg] | 84 (9) | 90 (7) | 89 (7) | 88 (8)
Potassium [Mean (Standard Deviation); unit: mmol/L] | 3.36 (0.45) | 3.55 (0.31) | 3.54 (0.41) | 3.49 (0.39)
24-hour Urinary Tetrahydroaldosterone Content (uTHA) [Median (Inter-Quartile Range); unit: ug/24h] | 80.0 [54.0 to 102.0] | 59.5 [41.0 to 76.0] | 69.0 [56.0 to 76.0] | 67.0 [45.0 to 97.0]

OUTCOME MEASURES:

1. Primary Outcome: Change in Aldosterone-to-renin Ratio
Description: Change from baseline in aldosterone-to-renin ratio (ARR) after 8 weeks of dexfadrostat phosphate treatment by dose group.
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: ng*L/dL*mU
Groups:
- 4 mg DP13; 8 mg DP13; 12 mg DP13; All Dose Arms Combined: Values are after 8 weeks of treatment with dexfadrostat phosphate
Arm/Group | 4 mg DP13 | 8 mg DP13 | 12 mg DP13 | All Dose Arms Combined
Number analyzed (Participants) | 10 | 12 | 13 | 35
ng*L/dL*mU | -15.0 [-25.5 to -5.7] | -7.0 [-16.0 to -2.7] | -14.0 [-20.8 to -8.4] | -11.8 [-23.8 to -4.9]
Statistical Analysis 1: Comparison: 4 mg DP13; Test type: Superiority; p < 0.0001, Mixed Models Analysis — The threshold value for statistical significance was p<0.05

2. Primary Outcome: Change in Ambulatory Systolic Blood Pressure
Description: All patients receiving at least one dose of dexfadrostat phosphate; analysis of all dose arms combined.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | 4 mg DP13 | 8 mg DP13 | 12 mg DP13 | All Dose Arms Combined
Number analyzed (Participants) | 10 | 12 | 13 | 35
mm Hg | -8 (10) | -14 (8) | -10 (9) | -11 (9)
Statistical Analysis 1: Comparison: 4 mg DP13; Test type: Superiority; p < 0.0001, Mixed Models Analysis — The threshold for significance was p <0.05

3. Secondary Outcome: Change in Potassium
Description: Change from baseline after 8 weeks of treatment with dexfadrostat phosphate
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | 4 mg DP13 | 8 mg DP13 | 12 mg DP13
Number analyzed (Participants) | 10 | 12 | 13
mmol/L | 0.74 (0.51) | 0.55 (0.29) | 0.28 (0.55)
Statistical Analysis 1: Comparison: 4 mg DP13; Test type: Superiority; p < 0.0001, Mixed Models Analysis — The threshold for significance was p <0.05

4. Secondary Outcome: Change in Ambulatory Diastolic Blood Pressure
Description: Change from baseline following 8-weeks of dexfadrostat phosphate treatment
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | 4 mg DP13 | 8 mg DP13 | 12 mg DP13
Number analyzed (Participants) | 10 | 12 | 13
mm Hg | -4.5 (7.0) | -7.9 (6.4) | -4.5 (7.0)
Statistical Analysis 1: Comparison: 4 mg DP13; Test type: Superiority; p < 0.0001, Mixed Models Analysis — The threshold for significance was p <0.05

5. Secondary Outcome: Change in 24-hour Urinary Tetrahydroaldosterone Content (uTHA)
Description: Change from baseline in urinary tetrahydroaldosterone content (uTHA) following 8 weeks of treatment with dexfadrostat phosphate
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: ug/24 hour urine
Groups:
- 4 mg DP13; 8 mg DP13; 12 mg DP13: Values are 8 weeks of treatment with dexfadrostat phosphate
Arm/Group | 4 mg DP13 | 8 mg DP13 | 12 mg DP13
Number analyzed (Participants) | 10 | 12 | 13
ug/24 hour urine | -61.0 [-86.0 to -45.0] | -50.0 [-74.0 to -28.5] | -66.0 [-71.0 to -41.0]
Statistical Analysis 1: Comparison: 4 mg DP13; Test type: Superiority; p < 0.0001, Mixed Models Analysis — The statistical threshold was p<0.05

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline (before treatment with dexfadrostat phosphate) to the end of 8 weeks of treatment with dexfadrostat phosphate
Description: All patients receiving at least one dose of dexfadrostat phosphate (safety population). The safety population included the full analysis set.
Groups:
- 4 mg DP13: Patients receiving low dose dexfadrostat phosphate daily for 8 weeks
- 8 mg DP13: Patients receiving middle dose dexfadrostat phosphate daily for 8 weeks
- 12 mg DP13: Patients receiving high dose dexfadrostat phosphate daily for 8 weeks
Arm/Group | 4 mg DP13 | 8 mg DP13 | 12 mg DP13
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 4/10 | 6/12 | 7/13
OTHER ADVERSE EVENTS (reported when occurring in more than 2.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4 mg DP13 (N=10) | 8 mg DP13 (N=12) | 12 mg DP13 (N=13)
Amylase increase (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increase (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood pressure diastolic increase (Investigations) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (4) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Polymenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Dyspnea during exercise
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower limb edema (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-12): https://cdn.clinicaltrials.gov/large-docs/06/NCT04007406/Prot_SAP_000.pdf